CLINICAL TRIAL: NCT07038070
Title: A Randomized Controlled Trial Comparing the Efficacy of Topical Vaginal Estrogen Versus Topical Vaginal Estrogen Plus Via, a Hyaluronic Acid-Based Vaginal Moisturizer, in the Treatment of Genitourinary Syndrome of Menopause
Brief Title: Via, a Hyaluronic Acid (HLA) Based Vaginal Moisturizer Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 25-00415
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Genitourinary Syndrome of Menopause (GSM)

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Vaginal Estrogen + Hyaluronic acid (HLA) (Experimental): Participants will administer vaginal estrogen tablets nightly for 2 weeks, then twice weekly for 14 weeks. Participants will concomitantly apply Via (Hyaluronic acid) nightly for 16 weeks.
  Interventions: Drug: Vaginal estrogen tablet; Device: Via Solv Wellness (Hyaluronic Acid Therapy)
- Vaginal Estrogen Alone (Active Comparator): Participants will administer vaginal estrogen tablets nightly for 2 weeks, then twice weekly for 14 weeks.
  Interventions: Drug: Vaginal estrogen tablet

INTERVENTIONS:
Drug: Vaginal estrogen tablet — The dosage of the vaginal estrogen will be one 10mcg tablet administered vaginally nightly for 2 weeks, then administered vaginally twice weekly for 14 weeks.
Device: Via Solv Wellness (Hyaluronic Acid Therapy) — The dosage of Via will be a pea-sized amount applied vaginally along the vaginal and vulvar walls nightly for 16 weeks.
  Arms: Vaginal Estrogen + Hyaluronic acid (HLA)

SUMMARY:
This study aims to evaluate whether the administration of vaginal estrogen along with Via, a hyaluronic acid-based vaginal moisturizer, offers superior relief from symptoms of genitourinary syndrome of menopause (GSM) in the urogynecologic patient population, compared to administration of vaginal estrogen alone.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal (last menstrual period at least 12 months ago).
* Aged 45 years or older and have symptoms of Genitourinary Syndrome of Menopause (GSM).
* Have never tried vaginal estrogen therapy, or have tried vaginal estrogen therapy, but have not used vaginal estrogen and/or hyaluronic acid products for management of GSM symptoms within the last 3 months.
* Capable of signing informed consent.
* Capable and willing to follow all study-relation visits.

Exclusion Criteria:

* Subjects currently diagnosed with or undergoing treatment for hormone-sensitive disease (e.g. breast cancer)
* Subjects currently using systemic hormone replacement therapy
* Subjects currently using estrogen hormonal therapies or hormone modulators (aromatase inhibitors or selective estrogen receptor modulators)

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Percent change in vulvovaginal symptom questionnaire (VSQ) score | Baseline, Week 16
  The VSQ is a 21-item survey designed to measure vaginal symptoms, emotions, life impact due to vulvovaginal symptoms, and sexual impact of vulvovaginal symptoms. The scores range from 0 - 20 with the higher score meaning greater impact from vulvovaginal symptoms.

SECONDARY OUTCOMES:
Percent change in vaginal pH | Baseline, Week 16
Change in vaginal maturation index (VMI) | Baseline, Week 16
  The number of parabasal cells, intermediate cells, and superficial cells will be counted, and the maturation index will be calculated as the percent basal cells visualized.
Number of adverse events related to treatment | Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Brucker, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared upon reasonable request beginning 9 to 36 months after publication or as required by a condition of awards or supporting agreements, provided the requesting investigator executes a data use agreement with NYU Langone Health. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's Data Sharing Strategy Board (DSSB). Requests should be directed to benajmin.brucker@nyulangone.org. The protocol and statistical analysis plan will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to benajmin.brucker@nyulangone.org. To gain access, data requestors will need to sign a data access agreement. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's DSSB.